CLINICAL TRIAL: NCT01536964
Title: The Effect of Morphine on Prasugrel Absorption in STEMI Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STH16207; 2011-003320-12 (EudraCT Number)
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Morphine; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Morphine (Experimental): the effect of morphine on prasugrel absorption will be tested
  Interventions: Drug: morphine
- Saline (Placebo Comparator)
  Interventions: Drug: saline

INTERVENTIONS:
Drug: morphine — 2.5mg of morphine will be given post Prasugrel administration with a further 2.5mg 5 minutes later
  Arms: Morphine
Drug: saline — 2.5ml of saline will be given post Prasugrel followed by a further 2.5ml as a comparator for the morphine
  Arms: Saline

SUMMARY:
Heart Attacks are a major cause of death in this country. When patients have a heart attack, they are treated with anti-clotting drugs, one of which is a drug called Prasugrel. It is important that Prasugrel starts to work as quickly as possible following a heart attack. As many patients who have a heart attack experience excruciating pain, they are often given morphine (a strong painkiller) by the Ambulance crew. We think that morphine may affect how Prasugrel is absorbed from the stomach and may delay how quickly it starts to work. We intend to study the effect of morphine on the absorption of Prasugrel.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age and willing and able to provide informed consent
* Admission to hospital with a STEMI >12 months prior to recruitment
* Previous prasugrel and morphine use with no adverse effect

Exclusion Criteria:

* Active respiratory disorder, resting oxygen saturation < 95% or decompensated congestive cardiac failure
* Current use of anti-platelet or anti-coagulant drugs apart from aspirin 75 mg daily, or receipt of any dose of clopidogrel, prasugrel or ticagrelor in the last 2 weeks
* Current use of opiate analgesia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
VerifyNow P2Y12 PRU measurement at 2 hours post dose | 2 hours
  Assessment of platelet function

SECONDARY OUTCOMES:
Estimated time to PRU less than 150; maximal LTA response to ADP 20 microM at 2 hours post dose; final LTA response to ADP 5 microM at 2 hours post dose. | 2 hours
  further assessment of platelet function

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom